CLINICAL TRIAL: NCT01161355
Title: An Exploratory Study to Assess the Absolute Bioavailability of a Single Oral Dose of AZD9668 With Respect to an Intra-venous Microdose of [14C]AZD9668 in Healthy Male Subjects
Brief Title: Phase I, Exploratory, Single Centre, Single Oral Dose AZD9668 and Intravenous Microdose of [C14] AZD9668, Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0520C00021
Record Dates: First submitted 2010-06-18; First posted 2010-07-13 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Safety; tolerability; healthy; microdose
MeSH Terms: interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9668 (Experimental): Tablets and intravenous (IV) dose
  Interventions: Drug: AZD9668

INTERVENTIONS:
Drug: AZD9668 — Tablets of AZD9668 and IV dose of [C14]AZD9668

SUMMARY:
The primary objective of this study is to assess the absolute bioavailability and to evaluate pharmacokinetic parameters of a single oral dose and a radiolabelled intravenous microdose of [14C]AZD9668 in healthy male subjects.

DETAILED DESCRIPTION:
This is an exploratory study to assess the absolute bioavailability of a single oral dose of AZD9668 with respect to an intra-venous microdose of [14C]AZD9668 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weight at least 50 kg and no more than 100 kg.

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically significant abnormalities at screening examination

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The absolute bioavailability and evaluation of pharmacokinetic parameters (AUC, AUC (0-t), Cmax, t½, tmax, and MRT of of a single oral dose and a radiolabelled intravenous microdose of [14C]AZD9668 | Multiple Pharmacokinetic blood samples for up to 96 hours following drug administration

SECONDARY OUTCOMES:
Safety and tolerability of AZD9668: Adverse events, clinical chemistry, haematology, urinalysis, vital signs, electrocardiogram, physical examination | measured within 21 days of drug administration and up to 7 days following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Marks-Konczalik, Study Director — AstraZeneca; Sharan Sidhu, MB ChB, BAO,, Principal Investigator — Quintiles, Inc.
Locations (2):
- United Kingdom (2):
  - Research Site, Ruddington, Nottingham
  - Research Site, London